CLINICAL TRIAL: NCT07245316
Title: Avoiding Surgery in Estrogen Receptor Positive Atypical Ductal Hyperplasia and In-situ Carcinoma Treated With Endocrine Treatment Trial
Acronym: ASAIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jeong Eon Lee (Other)
Responsible Party: Sponsor-Investigator, Jeong Eon Lee, Professor, Department of Surgery, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2025-02-036
Record Dates: First submitted 2025-08-20; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Ductal Carcinoma in Situ of the Breast
Keywords: ASAIN
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active monitoring arm (Experimental): Active monitoring with endocrine therapy in hormone-receptor positive, HER-2 negative DCIS, LCIS, ADH without surgery
  Interventions: Procedure: Avoiding surgery

INTERVENTIONS:
Procedure: Avoiding surgery — Avoiding surgery in hormone-receptor positive atypical ductal hyperplasia and in-situ carcinoma treated with endocrine treatment

SUMMARY:
This study aims to evaluate the 5-year invasive ipsilateral breast cancer incidence rate in patients with hormone-receptor positive, HER-2 negative atypical ductal hyperplasia or in-situ carcimona who omitted surgery and received endocrine therapy.

ELIGIBILITY:
1. Inclusion criteria:

1. Female patients aged ≥35 years.
2. Diagnosed with atypical ductal hyperplasia (ADH), ductal carcinoma in situ (DCIS), or lobular carcinoma in situ (LCIS) on core-needle biopsy, vacuum-assisted biopsy, or excisional biopsy.
3. Immunohistochemistry (IHC) performed on biopsy specimens confirming estrogen receptor (ER), progesterone receptor (PR), and HER2 status; eligible only if the ER Allred total score is ≥7 and HER2 status is negative.
4. All low- and intermediate-grade nuclear grades included; for high-grade lesions, only patients with a Ki-67 index ≤20% are eligible.
5. Lesion not definitely palpable on physical examination at diagnosis.
6. No prior breast surgery for ipsilateral or contralateral breast cancer, and no synchronous contralateral breast cancer.
7. Not diagnosed with pregnancy-associated breast cancer or breast cancer detected during lactation.
8. Negative serum or urine β-hCG prior to enrollment.
9. Provided written informed consent to participate in the study.

2. Exclusion criteria:

1. Pregnant patients.
2. Patients with clinically significant psychiatric disorders (e.g., major depressive disorder) or those currently receiving psychiatric or antipsychotic medications.
3. Concomitant diagnosis of invasive breast cancer.
4. Evidence of axillary lymph node metastasis.
5. Carriers of BRCA1/2 mutations.
6. Male patients.
7. History of diagnosis or treatment for breast cancer.
8. Presence or history of other malignancies besides breast cancer.
9. Concomitant diagnosis of pleomorphic LCIS.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
5 year ipsilateral breast cancer incidence rate | 5 years after the last patient enrollment
  This study aims to evaluate the 5-year invasive ipsilateral breast cancer incidence rate in patients with hormone-receptor positive, HER-2 negative atypical ductal hyperplasia or in-situ carcimona who omitted surgery and received endocrine therapy.

SECONDARY OUTCOMES:
Adjuvant chemotherapy rate | 5 years after the last patient enrollment
  5 year adjuvant chemotherapy rate
invasive CBC rate | 5 years after the last patient enrollment
  5 year invasive contralateral breast cancer rate
OS | 5 years after the last patient enrollment
  5 year overall survival
BCSS | 5 years after the last patient enrollment
  5 year breast cancer specific survival
Change in health-related quality of life assessed by EORTC QLQ-C30 | At baseline, at 2 years, and at 5 years after the last patient enrollment
  HRQoL will be evaluated using the EORTC QLQ-C30. Scores range from 0-100. Higher functional/global health scores indicate better QoL, while higher symptom scores indicate greater symptom burden.
Change in breast cancer-specific quality of life assessed by EORTC QLQ-BR23 | At baseline, at 2 years, and at 5 years after the last patient enrollment
  Breast cancer-specific QoL will be assessed using the EORTC QLQ-BR23. Scores range from 0-100. Higher functional scores indicate better QoL; higher symptom scores indicate worse symptom burden.

OTHER OUTCOMES:
Prognostic differences in invasive breast cancer progression according to age and type of endocrine therapy | 5 years after the last patient enrollment
  Invasive breast cancer progression will be evaluated according to age at diagnosis and type of endocrine therapy. The proportion of participants who develop histologically confirmed invasive breast cancer during follow-up will be compared across subgroups defined by age and endocrine therapy regimen (tamoxifen, aromatase inhibitor, or combination with ovarian function suppression).
Adverse events associated with endocrine therapy and ovarian function suppression | From initiation of endocrine therapy to treatment discontinuation or last follow-up (up to 5 years after enrollment)
  Incidence and severity of adverse events related to endocrine therapy and/or ovarian function suppression, graded according to CTCAE criteria.
Direct medical cost of active monitoring compared with standard therapy | 5 years after the last patient enrollment
  Mean total direct medical cost (USD) incurred during 5-year follow-up will be compared between the active monitoring protocol and standard surgical management based on institutional billing data.
Incremental cost-effectiveness ratio (ICER) of active monitoring compared with standard therapy | 5 years after last patient enrollment.
  Cost-effectiveness will be evaluated by the incremental cost-effectiveness ratio (ICER), calculated as cost per quality-adjusted life-year (QALY) gained for active monitoring versus standard therapy.
Change in circulating tumor DNA (ctDNA) detectability from baseline to surgery among participants who undergo surgery for invasive progression | Baseline and at time of surgery
  Paired assessment of ctDNA detectability (present/absent) at baseline (diagnosis) and at the time of surgery among participants who progress to invasive breast cancer. Peripheral blood (20 mL) is collected at both time points.
Longitudinal detectability of circulating tumor DNA (ctDNA) at annual follow-up compared with baseline | Baseline (Day 1) and annually through study completion (up to 5 years)
  Assessment of ctDNA detectability (present/absent) at baseline and at annual follow-up visits in all enrolled participants. Peripheral blood (20 mL) is collected at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Eon Lee, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No